CLINICAL TRIAL: NCT06441656
Title: The (Flip and Fix) Internal Limiting Flap Technique Versus the Classic Temporal Flap for Macular Hole Repair
Acronym: Flip and Fix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Islam Shereen Hamdy, Associate Professor, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Flip and Fix ILM flap
Record Dates: First submitted 2024-05-29; First posted 2024-06-04 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-05

CONDITIONS: Hacular Hole Repair
Keywords: Macular hole, Internal limiting membrane, pars plana vitrectomy, perfluorocarbon liquid, non-heparinized blood
MeSH Terms: conditions — Retinal Perforations | interventions — Vitrectomy

STUDY DESIGN:
Intervention Model Description: Prospective comparative
Who Masked: Participant, Care Provider, Outcomes Assessor
Masking Description: The investigator assessing the outcome was masked to the type of surgery done
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Flip and fix ILM flap (Experimental): In the (Flip and Fix) technique group, the (flipped) ILM flap was secured in place and flattened over the macular surface using a 1.5 cc bubble of PFCL (Arcaline; Arcadophtha, Toulouse, France) injected over the flipped ILM flap. Then fluid air exchange with removal of the PFCL bubble was done followed by (fixing) the ILM flap over the macular surface using two drops of autologous non-heparinized blood -collected by the attending nurse or anaesthesiologist from one of the veins on the dorsum of the hand- one dropped over the superior-nasal and another at the inferior-nasal edges of the ILM flap (away from the MH center).
  Interventions: Procedure: Vitrectomy with ILM flap
- classic temporal ILM flap (Active Comparator): PFCL and blood were not used to fix the ILM flap
  Interventions: Procedure: Vitrectomy with ILM flap

INTERVENTIONS:
Procedure: Vitrectomy with ILM flap — In both groups, a single-layer ILM temporal flap of approximately 2 times the size of the optic disc was fashioned using an ILM forceps temporal to the macula. The nasal edge of the flap was not detached from the temporal MH edge. The flap was reflected nasally to cover the MH

SUMMARY:
Purpose To describe a novel technique of MH repair and compare it to the perfluorocarbon liquid (PFCL) assisted temporal ILM flap technique.

Methods Twenty-two eyes of 22 patients with MH were randomized on 1:1 basis into two groups. Group A cases were treated using the (Flip and Fix) technique in which the single-layer ILM flap was (flipped), flattened over the macula using PFCL and (fixed) in place using 2 drops of autologous non-heparinized blood over the superonasal and the inferonasal edges of the flap (away from the MH center). Group B patients had the classic temporal ILM flap technique without using the PFCL or autologous blood. All patients were followed up for a period of 6 months after the surgery.

Results No significant difference was observed in initial and final visual acuities between Groups A and B. Intraoperative flap displacement and did not occur in Group A and occurred in 2 eyes in Group B (18.2%) one of them showed failed MH closure and required reoperation, These 2 cases had a final (W shape) MH closure and a worse final vision than the remaining cases which had either (U shape) or (V shape) final MH closure.

Conclusions The study results show that the (Flip and Fix) technique is as effective as the PFCL-assisted temporal ILM flap technique and is associated with less ILM flap displacement risk for the repair of macular holes.

DETAILED DESCRIPTION:
We conducted a prospective randomized comparative interventional study in which we enrolled patients older than 50 years with idiopathic macular holes who presented to (Removed in the blinded version of manuscript) in the period between February 2021 and February 2022. Patients with previous macular surgeries and those with any other significant macular pathologies e.g., diabetic macular oedema, myopic maculopathy, choroidal neovascular membrane, or macula-off retinal detachment were excluded.

The study protocol was reviewed and approved by the Ethics Committee of (Removed in the blinded version of manuscript). All patients signed an informed consent after explaining the procedures. The study was conducted in accordance with the tenets of the Declaration of Helsinki.

For all the patients, a retina consultant (I. A.) masked to the procedure that will be done for the patient conducted a comprehensive ophthalmic examination, including best-corrected visual acuity (BCVA) (measured using the Snellen's chart and then converted to the LogMAR for the statistical analysis), slit-lamp examination, and fundus examination.

All the patients had a pre-operative macular OCT scan done. The scans were assessed by the masked retina consultant (I. A.) to confirm the diagnosis and to measure the minimum MH diameter.

The included patients were randomized by a research nurse on a 1:1 basis using the closed envelope technique to have either the new (Flip and fix) technique (Group A) or the PFCL assisted temporal inverted ILM flap technique (Group B).

All the surgeries were done under general anaesthesia by a single surgeon (M. A.) using a wide-angle viewing non-contact system (Resight; Carl Zeiss Meditec AG, Jena, Germany) and 23 Gauge Alcon Constellation vitrectomy machine (Alcon Laboratories, Fort Worth, TX) to complete the core vitrectomy and induction of the posterior vitreous detachment if not already detached, this was followed by an injection the Brilliant Blue G (Tissueblue 0.025% DORC, Zuidland, The Netherland) to stain the ILM.

In both groups, a single-layer ILM temporal flap of approximately 2 times the size of the optic disc was fashioned using an ILM forceps temporal to the macula. The nasal edge of the flap was not detached from the temporal MH edge. The flap was reflected nasally to cover the MH In the (Flip and Fix) technique group, the (flipped) ILM flap was secured in place and flattened over the macular surface using a 1.5 cc bubble of PFCL (Arcaline; Arcadophtha, Toulouse, France) injected over the flipped ILM flap. Then fluid air exchange with removal of the PFCL bubble was done followed by (fixing) the ILM flap over the macular surface using two drops of autologous non-heparinized blood -collected by the attending nurse or anaesthesiologist from one of the veins on the dorsum of the hand- one dropped over the superior-nasal and another at the inferior-nasal edges of the ILM flap (away from the MH center). On the other hand, in the classic temporal ILM flap group, PFCL and blood were not used to fix the ILM flap. Videos demonstrating the technique are provided as supplemental files 1 and 2.

In both groups, at the conclusion of the surgery the air was exchanged for a non-expansile concentration (20%) of sulphur hexafluoride gas SF6 and the patient was asked to maintain a face -down position for 5 days postoperatively. The surgical steps of the (flap and fix) technique are summarized in Figure 1.

For all the cases, intraoperative ILM flap displacement (defined as a significant displacement of the inverted ILM flap after its initial positioning over the MH that necessitated readjustment) was reported by the operating surgeon.

All the patients were examined postoperatively at 1, 3, and 6 months by a retina consultant masked to the used surgical procedure (I. A). The best corrected visual acuity, slit-lamp examination, fundus examination and macular OCT scanning were done in each postoperative visit.

According to the cross-sectional morphology on the postoperative macular OCT scan, foveal contour was classified into one of the following categories: U-shape, V-shape, and W-shape (irregular). The presence of a thin hyperreflective band of tissue extending on both sides of the previous MH Flap between the inner surface of the retina was assessed and considered a (membranous i.e., flap closure).

The data about the pre-operative MH base size, minimum MH diameter, BCVA, post-operative closure rate, BCVA, and the pattern of the MH closure was collected.

ELIGIBILITY:
Inclusion Criteria: patients with idiopathic macular holes who presented to (Removed in the blinded version of manuscript) in the period between February 2021 and February 2022.

Exclusion Criteria: Patients with previous macular surgeries and those with any other significant macular pathologies e.g., diabetic macular oedema, myopic maculopathy, choroidal neovascular membrane, or macula-off retinal detachment -

-

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2022-02-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
Macular hoe closure by OCT scan | 1, 3, and six months postoperatively
  Macular OCT scan was used to assess the MH closure
LogMAR visual acuity | 1, 3, and six months postoperatively
  Best corrected visual acuity was assessed using the LogMAR vision

CONTACTS AND LOCATIONS:
Overall Officials: Islam SH Ahmed, M.D., Principal Investigator — University of Alexandria
Locations (1):
- Faculty of Medicine Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No
The data are available upon request